CLINICAL TRIAL: NCT07226687
Title: A Randomized Controlled Trial Evaluating the Impact of Small Versus Large Urethral Bites on Continence Outcomes After Robotic Radical Prostatectomy
Brief Title: Evaluating the Impact of Small Versus Large Urethral Stiches (or 'Bites') on Urinary Continence.
Acronym: STITCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB25-0202
Record Dates: First submitted 2025-09-23; First posted 2025-11-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Prostatectomy
Keywords: Prostatectomy; Urinary continence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Bites (Experimental): Patients will undergo Robotic-assisted radical prostatectomy (RARP) with vesicourethral anastomosis using small urethral bites, as determined by the surgeon, with goal of being approximately 5-7 mm from the cut edge of the urethra.
  Interventions: Procedure: Small Urethral Bite Technique
- Large Bites (Experimental): Patients will undergo Robotic-assisted radical prostatectomy (RARP) with vesicourethral anastomosis using large urethral bites, as determined by the surgeon, with goal of being approximately 15-20 mm from the cut edge of the urethra.
  Interventions: Procedure: Large Urethral Bite Technique

INTERVENTIONS:
Procedure: Small Urethral Bite Technique — The small urethral bite technique involves placing sutures (stitches) that are ~5-7 mm from the edge of the urethra. Each suture penetrates the full thickness of the urethra.
  Arms: Small Bites
Procedure: Large Urethral Bite Technique — The large urethral bite technique involves placing sutures (stitches) that are ~15-20 mm from the edge of the urethra. Each suture penetrates the full thickness of the urethra.
  Arms: Large Bites

SUMMARY:
To evaluate the impact of sustainable functional urethral reconstruction (SFUR) on early recovery of urinary continence (UC) after robot-assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years and older.
* Diagnosis of prostate cancer with an indication for robotic-assisted radical prostatectomy (RARP).
* Ability to provide informed consent.

Exclusion Criteria:

* History of pelvic radiation therapy
* Prostatectomy performed in the context of salvage therapy (e.g., post-radiation or post-focal therapy)
* Presence of extra-pelvic metastatic disease
* Neurological disorders significantly affecting continence (e.g., severe Parkinson's disease, multiple sclerosis)
* Pre-existing urinary incontinence
* Inability to comply with follow-up protocols

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2031-05-23 (Estimated); Study Completion 2031-05-23 (Estimated)

PRIMARY OUTCOMES:
Evaluating the impact of the urethral bites | 6 months following RARP
  To evaluate the impact of small versus large urethral bites during vesicourethral anastomosis on urinary continence at 6 months following Robotic-assisted radical prostatectomy (RARP). Specifically, we aim to determine whether a smaller or larger suture bite technique results in superior continence recovery. This will be measured by comparing the number of incontinence pads that are needed to be used per day between each group.

SECONDARY OUTCOMES:
Assessment of urinary leaks and complications | 3 months following surgery
  Assessing the rate of anastomotic urinary leaks and overall surgical complication rates.
Assessment of urinary leaks and complications | 12 months following surgery
  Assessing the rate of anastomotic urinary leaks and overall surgical complication rates.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Eggener, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States